CLINICAL TRIAL: NCT05750342
Title: Randomized Clinical Trial to Analyze the Efficacy of a Supplement Extracted From Persimmon on Overweight / Obesity Grade I in Subjects With Body Mass Index Greater Than 25.
Brief Title: Clinical Trial to Analyze the Efficacy of a Supplement Extracted From Persimmon on Overweight / Obesity.
Acronym: PERSOB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Francisco Javier López Román, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: UCAMCFE-00032
Record Dates: First submitted 2023-01-30; First posted 2023-03-01 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2023-01

CONDITIONS: Supplementation; Obesity
Keywords: Obesity; Overweight; Persimmon
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caqui (Experimental): Subjects will consume two capsules daily. Each capsule will be taken before the two main meals.
  Interventions: Dietary Supplement: Experimental Product Caqui
- Placebo (Placebo Comparator): The product will have the same characteristics as the experimental product. They will consume two capsules per day, one before the two main meals.
  Interventions: Dietary Supplement: Control product placebo

INTERVENTIONS:
Dietary Supplement: Experimental Product Caqui — Supplement extracted from persimmon
  Arms: Caqui
Dietary Supplement: Control product placebo — Product with identical characteristics to the experimental product.
  Arms: Placebo

SUMMARY:
Randomized, controlled, double-blind clinical trial, with two parallel branches depending on the product consumed (experimental product and placebo product) and single-center, to measure the efficacy of a supplement extracted from Persimmon on overweight and obesity grade I in subjects with BMI over 25.

DETAILED DESCRIPTION:
The product to be consumed is a supplement extracted from the Persimmon. Participants will consume the product for 84 days. They will take one capsule before the two main meals.

Subjects will have to make 3 visits to the laboratory. In the initial visit it will be verified if the subject meets the criteria required by the study. Subjects who meet the selection criteria will be randomly assigned to each of the study groups (investigational product or placebo, depending on the group to which they have been assigned).

In the other two visits, the subjects will carry out the appropriate tests for taking of data colletion. These visits will be separated by 84 days of product consumption.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of both sexes aged 18-65 years.
* Subjects with a body mass index greater than 25 and less than 35.
* Volunteers able to understand the clinical study and willing to comply with the study procedures and the procedures and requirements of the study.

Exclusion Criteria:

* Subjects undergoing treatment that may affect body weight.
* Subjects with acute diseases.
* Volunteers with a history or presence of chronic pulmonary disorders, hepatic, renal, hematological, gastrointestinal, endocrine, immunological, dermatological, urological, neurological, psychiatric, cardiovascular, or malignant tumor pathology or disease.
* Subjects who have undergone major surgery in the last 3 months.
* Subjects who quit smoking in the last 6 months or who intend to quit during the study.
* Subjects with allergies or eating disorders.
* Volunteers who are participating in another study that involves blood draws or dietary intervention.
* Pregnant or breastfeeding women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-05-06 (Actual)

PRIMARY OUTCOMES:
Total fat mass | From baseline to 84 days
  Dual X-ray absorptiometry (DEXA), measured in grams.
Fat mass in torso | From baseline to 84 days
  Dual X-ray absorptiometry (DEXA), measured in grams.
Fat mass in lower limbs | From baseline to 84 days
  Dual X-ray absorptiometry (DEXA), measured in grams.

SECONDARY OUTCOMES:
Fat mass | A record of body composition will be made twotimes during the 84 days of consumption. Measures will be taken at baseline, and at 84 days. For this we will use a TANITA.
  body composition measured by bioimpedancemetry
Muscle mass | A record of body composition will be made twotimes during the 84 days of consumption. Measures will be taken at baseline, and at 84 days. For this we will use a TANITA.
  body composition measured by bioimpedancemetry
Percentage of fat mass | A record of body composition will be made twotimes during the 84 days of consumption. Measures will be taken at baseline, and at 84 days. For this we will use a TANITA.
  body composition measured by bioimpedancemetry
Waist-hip perimeter | A record of body composition will be made twotimes during the 84 days of consumption. Measures will be taken at baseline, and at 84 days. For this we will use a TANITA.
  The waist and hips will be measured, in centimeters.
Lipidic Metabolism | Blood samples will be taken twice, once at baseline, at the beginning of the trial and once at the end after 84 days of product intake.
  Total cholesterol, LDL, oxidized LDL, HDL, and triglycerides. Will be measured in milligrams per deciliter.
Glycidic profile | Blood samples will be taken twice, once at baseline, at the beginning of the trial and once at the end after 84 days of product intake.
  Blood glucose, glycated hemoglobin and basal insulin. It was measured in milligrams per deciliter.
Quality of life in people with obesity | The questionnaire will be carried out twice. The first time at the beginning and the second after carrying out 84 days of consumption of the product under study.
  Assessed using the Obesity and Quality of Life Consulting test (IWQol-Lite)
Total antioxidant capacity of plasma | Blood samples will be taken twice, once at baseline, at the beginning of the trial and once at the end after 84 days of product intake.
  It will be done through the OxiSelect Total Antioxidant Capacity (TAC) Assay Kit
Inflammatory profile - PCR | Blood samples will be taken twice, once at baseline, at the beginning of the trial and once at the end after 84 days of product intake.
  C-Reactive Protein will be measured
Inflammatory profile - IL-6 | Blood samples will be taken twice, once at baseline, at the beginning of the trial and once at the end after 84 days of product intake.
  Interlucin 6 will be measured
Gut microbiota | Stool collection will be performed twice on subjects. The first time at the beginning and the second after 84 days of consumption of the product under study.
  Evaluated with stool sample
Physical activity | An accelerometer will be placed twice on the subjects. The first time at baseline and the second after taking 84 days of consumption of the product under study
  Measured with Actigraph wGT3X-BT
Nutritional assessment | The food recall will be performed twice on the subjects. The first time at the beginning and the second after carrying out 84 days of consumption of the product under study. In each one a total of 7 days will be collected.
  "24-hour recall" food survey.
Liver safety variables | Hematological samples were taken before (day 0) and after consumption of the product (day 84) both in the control group and in the experimental group.
  It is a blood test that measures the presence of some enzymes, proteins and bilirubin in the blood, with the aim of determining if there is any alteration in the liver. Enzyme GPT, GOT, Gamma GT, LDH, alkaline phosphatase and bilirubin (UI/L)

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Murcia, Murcia, Spain

REFERENCES:
- [Derived] Perez-Pinero S, Munoz-Carrillo JC, Echepare-Taberna J, Herrera-Fernandez C, Munoz-Camara M, Avila-Gandia V, Lopez-Roman FJ. Efficacy of a Dietary Supplement Extracted from Persimmon (Diospyros kaki L.f.) in Overweight Healthy Adults: A Randomized, Double-Blind, Controlled Clinical Trial. Foods. 2024 Dec 17;13(24):4072. doi: 10.3390/foods13244072. PMID 39767014